CLINICAL TRIAL: NCT04185051
Title: A Double-blind, Randomized, Placebo Controlled, 4-week Study to Investigate the Effect of JNJ-67953964 on Gastric Mucosal Integrity in Healthy Male and Female Participants
Brief Title: A Study to Investigate the Effect of JNJ-67953964 on Gastric Mucosal Integrity in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108686; 67953964EDI1001 (Other: Janssen Research & Development, LLC); 2019-001864-31 (EudraCT Number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: JNJ-67953964 or Placebo (Experimental): Participants will receive JNJ-67953964 or matching placebo oral capsules once daily (QD) over 4 weeks (28 days).
  Interventions: Drug: JNJ-67953964; Drug: Placebo
- Cohort 2: JNJ-67953964 or Placebo (Experimental): Participants in this cohort will receive JNJ-67953964 only or will be randomly assigned to receive JNJ-67953964 or matching placebo.
  Interventions: Drug: JNJ-67953964; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-67953964 — Participants will receive JNJ-67953964 as oral capsules.
  Other Names: Cerecor (CERC)-501
Drug: Placebo — Participants will receive matching placebo oral capsules.

SUMMARY:
The main purpose of the study is to investigate the upper gastro-intestinal (GI)-related safety and tolerability in healthy participants by gastroscopy and gastric biopsies after treatment with 25 milligram (mg) JNJ-67953964 once daily (QD) over 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 30 kilograms per meter square (kg/m^2). Minimum body weight should be 50 kilogram (kg)
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Non-smokers (not smoked for 3 months prior to screening)
* A woman of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test before the first dose
* A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person until 90 days after receiving the last dose of study intervention

Exclusion Criteria:

* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* History of any gastric surgery, documented gastric disease (including peptic ulcer disease, gastritis, achlorhydria, upper gastro-intestinal (GI) bleeding, esophagitis, or any GI precancerous condition), current clinically evident GI complaints including functional gastrointestinal disorders (FGID)
* Is positive for helicobacter (H.) pylori antigen in a stool test at screening
* Is diagnosed to have any gastric disease (macroscopic) as visually assessed by gastroscopy at screening
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Microscopic Signs of Parietal Cell Damage | Day 28
  Microscopic signs of parietal cell damage is defined as the any of the following observations to be present in at least 2 biopsy specimens collected during a gastroscopy session: greater than (>) 25 percent (%) decrease in the number of parietal cells from baseline in the gastric biopsies at visit 4 or multifocal to diffuse parietal cell apoptosis or degeneration.

SECONDARY OUTCOMES:
Percentage of Participants with Microscopic Signs of Ulcers or Erosions in the Gastric Biopsies | Day 28
  Microscopic signs of ulcers or erosions in the gastric biopsies will be assessed by high resolution gastroscopy using the 5-point Lanza scale: 0 = normal stomach, 1= mucosal hemorrhages only, 2 = 1 or 2 erosions, 3 = numerous (3-10) areas of erosion, and 4 = large number of erosions (>10) or ulcer.
Percentage of Participants with a Gastroscopy Lanza Score Greater than or Equal to (>=) 2 | Day 28
  Gastroscopy lanza scale is a 5-point scale where: 0 = normal stomach, 1= mucosal hemorrhages only, 2 = 1 or 2 erosions, 3 = numerous (3-10) areas of erosion, and 4 = large number of erosions (>10) or ulcer.
Percentage of Participants with a Gastroscopy Lanza Score Equal to (=) 4 | Day 28
  Gastroscopy lanza scale is a 5-point scale where: 0 = normal stomach, 1= mucosal hemorrhages only, 2 = 1 or 2 erosions, 3 = numerous (3-10) areas of erosion, and 4 = large number of erosions (>10) or ulcer.
Distribution of all Gastroscopy Lanza Scores | Day 28
  Gastroscopy lanza scale is a 5-point scale where: 0 = normal stomach, 1= mucosal hemorrhages only, 2 = 1 or 2 erosions, 3 = numerous (3-10) areas of erosion, and 4 = large number of erosions (>10) or ulcer.
Gastric pH Before and up to 4 Hours After Dosing | Day 1: Predose up to 4 hours postdose
  Gastric pH before and up to 4 hours after dosing will be measured. To measure gastric pH a nasal-gastric tube will be placed about one hour before dosing and remain in place until 4 hours after dosing.
Percentage of Participants with Adverse Events (AEs) and AEs Related to Upper Gastrointestinal Symptoms | Up to 15 Weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency